CLINICAL TRIAL: NCT06056011
Title: TIMMY3 80601-2-56:2017 + A1 2018 Clinical Accuracy Study
Brief Title: Timmy3 Module Clinical Accuracy ISO 80601-2-56:2017 + A1 2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 60128116
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Febrile Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Oral Temperature Measurement (Experimental): Oral temperature measurements for subjects age Group C as 5 years or older. Both febrile and non-febrile subjects included in this arm.
  Interventions: Device: Connex CSVM with Timmy3 module
- Axillary Temperature Measurement (Experimental): Adult Axillary temperature measurement supports age Group C where C contains 18 years and older subjects.
  Pediatric Axillary temperature measurement supports newborn to 5 years and less than 18 years old.
  Both febrile and non-febrile subjects included in this arm.
  Interventions: Device: Connex CSVM with Timmy3 module
- Rectal Temperature Measurement (Experimental): Rectal temperature measurements for all age groups (newborn to subjects older than 18 years of age) with no restrictions. Both febrile and non-febrile subjects included in this arm.
  Interventions: Device: Connex CSVM with Timmy3 module

INTERVENTIONS:
Device: Connex CSVM with Timmy3 module — Connex Vital Signs Monitor with the Timmy3 Investigational module

SUMMARY:
The purpose of this document is to validate the clinical accuracy of the TIMMY3 thermometry module, integrated into host device CVSM, according to ISO 80601-2-56:2017 + A1 2018.

DETAILED DESCRIPTION:
The purpose of this document is to validate the clinical accuracy of the TIMMY3 thermometry module, integrated into host device CVSM, according to 80601-2-56:2017 + A1 2018.

This study is designed to provide supporting documentation for the TIMMY3 module operating with SureTemp Plus algorithms. Testing will be performed with a production equivalent CVSM modified to use TIMMY3 (TIMMY3 investigational device), running the SureTemp Plus algorithms. The TIMMY3 module is intended to be integrated into additional Welch Allyn devices such as, but not limited to, the Connex Spot Monitor and Spot 4400. The process described below will be followed in accordance with the method called out in ISO 80601-2-56:2017 + A1:2018.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects (person who is having their temperature taken) must meet the following criteria to participate in this study:

  * Subjects that are minors must provide assent to the clinical site's policy (if approved by Baxter) and/or the study sponsor's policy to participate in the study.
  * Subject or the legally authorized representative (LAR) must sign the informed consent form in order for the subject to participate.
  * Subject must be willing and able to comply with the study procedures.
  * Age: normal weight (full-term) newborn to adult
  * The study subject is in ambient temperature for at least 20 minutes prior to participating.
  * The study subject is able to have their temperature taken for up to six minutes for multiple rounds of temperatures per anatomical site.
  * The study subject is not physically or emotionally agitated/uncooperative.
  * The study subject or legal guardian speaks/understands fluent English.

Exclusion Criteria:

* Study subjects (person who is having their temperature taken) are excluded if they meet any of the below criteria. Any subject that withdraws from the study will be replaced.

  * The study subject has anatomical abnormalities that would affect temperature.
  * The study subject has any known contraindication to oral, axillary, or rectal temperature measurements.
  * The subject is not alert or unable to follow simple commands such as closing one's mouth completely around the probe if an oral reference temperature is being taken.
  * The study subject has consumed food or drink, or smoked, within the last 20 minutes. The subject may be included if they wait 20 minutes prior to taking oral temperature.
  * The study subject has engaged in strenuous or semi-strenuous activity within the last twenty minutes (i.e., running, weightlifting, etc.).
  * Subject has taken antipyretics (Aspirin, acetaminophen, ibuprofen) in the preceding 120 minutes.
  * Subjects has medical conditions such as inflammation at the MEASURING SITE (Barbiturates, thyroid preparations, antipsychotics, recent immunizations).
  * Neutropenic immunocompromised patients, in whom rectal manipulation may seed the blood with bacteria.

Note: The study subject will be excluded if the reference temperature does not stabilize after the 3 -5 minute monitoring time.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Validate the Clinical Accuracy of the Timmy3 thermometer algorithm | Up to 2 years
  All age groups in the oral, adult and pediatric axillary, and rectal temperature modes. Clinical accuracy will include measurement of clinical bias, with its limits of agreement, and clinical repeatability as defined by the ISO 80601-2-56:2017 + A1:2018.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fernandez, M.D., Study Director — Baxter Healthcare Corporation
Locations (5):
- United States (5):
  - First Georgia Physicians Group, Fayetteville, Georgia
  - Mankato Clinic, Mankato, Minnesota
  - John R. Oishei Children's Hospital, Buffalo, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Forest Lane Pediatrics, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No